CLINICAL TRIAL: NCT01533805
Title: Effects of Different Techniques of the Method Pilates in Chronic Low Back Pain in Women 46 to 60 Years
Brief Title: Effects of Different Techniques of the Method Pilates in Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Principal Investigator, Cintia Pereira de Souza, Principal Investigator, Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 0119031200011
Record Dates: First submitted 2012-02-02; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Low Back Pain
Keywords: Lumbago; Exercise therapy; Spine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilates with stabilization (Experimental): This group will do pilates exercises with a focus on control of segmental stabilization of the lumbar spine neutral.
  Interventions: Other: Pilates exercises with stabilization
- Classic Pilates (Active Comparator): This group will make Pilates exercises its focus is on mobilization exercises of the lumbar spine.
  Interventions: Other: Classic Pilates

INTERVENTIONS:
Other: Pilates exercises with stabilization — This group will focus on exercises with core stabilizing muscles. The frequency will be 16 sessions lasting 1 hour.
  Other Names: Pilates with stabilization segmental
  Arms: Pilates with stabilization
Other: Classic Pilates — This group will make Pilates exercises its focus is on mobilization exercises of the lumbar spine. The frequency will be 16 sessions lasting 1 hour.
  Arms: Classic Pilates

SUMMARY:
The purpose of this study is to compare different methods of application of the Pilates Method with exercises in controlling in low back pain in women aged between 45 and 60 years. Two groups will be formed. One will do Pilates exercises with stabilization segmental. The other group will do classic Pilates exercises. Will be measure pre and pos intervention of the responses already shown above.

DETAILED DESCRIPTION:
The purpose of this study is to identify what type of Pilates exercise is more effective in controlling low back pain is exercise that uses the method of the classical manner or trunk mobilizations with exercises that target the neutral position of the lumbar spine and deep muscles and focus on stabilizing the trunk.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain classified by visual analogue scale being 3-6 points to more than 3 weeks
* Not be performing any other type of physical therapy

Exclusion Criteria:

* Pregnant women
* Back surgeries
* Cardiovascular and rheumatic diseases

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain | Up to 8 weeks
  low back pain will be assessed with numeric pain scale two times (pre and post-intervention)

SECONDARY OUTCOMES:
Endurance of the back extensor muscles | Up to 8 weeks
  The endurance of the back extensor muscles will be assessed Biering-Sorensen test
Activity of abdominis transversus | Up to 8 weeks
  Will be assessed with Biofeedback pressure stabilizer
Functional Limitation | Up to 8 weeks
  Will be assessed Rolland Morris Test

CONTACTS AND LOCATIONS:
Overall Officials: Cintia P Souza, bachelor, Principal Investigator — University Gama Filho
Locations (1):
- Gama Filho University, Rio de Janeiro, Rio de Janeiro, Brazil